CLINICAL TRIAL: NCT04969640
Title: Role of Anterior Segment Optical Coherence Tomography in Staging and Evaluation of Treatment Response in Infectious Keratitis
Brief Title: Role of Anterior Segment Optical Coherence Tomography in Infectious Keratitis
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahemd Abdelghany, Assistant professor, Minia University
Other Study IDs: 43:6/2021
Record Dates: First submitted 2021-06-25; First posted 2021-07-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Infective Keratitis
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infective keratitis: 50 cases with infectious keratitis (any age) either received medical treatment or not, attending to our department will be included in the study.
  Interventions: Other: Optical coherence tomography

INTERVENTIONS:
Other: Optical coherence tomography — Anterior segment optical coherence tomography examination of corneas with infective keratitis

SUMMARY:
To evaluate the role of anterior segment optical coherence tomography in follow up of infectious keratitis and assessment of response to treatment.

DETAILED DESCRIPTION:
50 patients with proven infectious keratitis clinically will be included in the study.

The following will be performed for all patients in initial visit and follow up:

* Slit lamp examination and photography.
* Visual acuity assessment.
* Anterior segment optical coherence tomography.

  1. The central corneal thickness (CCT) (extracted from pachymetry map),
  2. Minimal corneal thickness (MCT) (extracted from pachymetry map)
  3. Corneal thickness at the site of the lesion (CTL) (extracted from pachymetry map or the sum of STL+ CETL)
  4. Stromal thickness at the center of the lesion (STL) stromal lesion (extracted from stromal map)
  5. Corneal epithelial thickness over the stromal lesion (CETL) at the center of the lesion (extracted from epithelial map)

ELIGIBILITY:
Inclusion Criteria:

* Any case with infectious keratitis (any age) either received medical treatment or not, attending to our department will be included in the study.

Exclusion Criteria:

* Cases with healed infectious keratitis.
* Cases presented from the start with severe corneal affection and melting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any case with infective keratitis
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
criteria of lesion on optical coherence tomography | 1 month
  Localiztion, depth of infiltration area in microns
width of lesion on optical coherence tomography | 1 month
  width of infiltration in microns

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelghany, ASS PROF, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided